CLINICAL TRIAL: NCT03937960
Title: Effect of Carbohydrate Restricted Versus Standard Low Fat Diet in the Treatment of Dyslipidemia in Children With Metabolic Syndrome
Brief Title: Effect of Low Carbohydrate Versus Low Fat Diet in the Treatment of Dyslipidemia in Obese Children With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Bhuvana Sunil, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300002816; P30DK056336 (NIH)
Record Dates: First submitted 2019-04-24; First posted 2019-05-06 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Metabolic Syndrome; Obesity; Dyslipidemias
Keywords: Dietary intervention; Anthropometric measure; Lipid profile; Augmentation Index; Flow mediated dilation; DXA scan; Nuclear magnetic resonance lipid profile
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate restricted group (Active Comparator): This diet is designed to minimize intake of carbohydrate sources such as added sugars, high glycemic grains, and fructose. It will provide a fixed amount of carbohydrate, and a total calorie goal - with proteins and fats to satiety. During the first two weeks of the intervention, carbohydrate (CHO) sources will be primarily derived from leafy greens and non-starchy vegetables and CHO intake will be equally distributed across meals throughout the day. At week three, additional CHO sources will be added back to the diet prescription including nuts, unsweetened yogurt, and low-glycemic fruits such as apples and berries.
  Interventions: Other: Carbohydrate restricted group
- Standard/Low fat diet group (Active Comparator): The control, low-fat diet will contain 55:25:20 %energy from CHO: protein: fat based on the United States Department of Agriculture (USDA) My Plate Daily Food Plan and our groups previous work. For example, an 1800 kcal/d plan will include 5 ounces lean meats, 3 cups low-fat dairy, 6 ounces of whole grains, 1 ½ cups fruit, 2 ½ cups vegetables (starchy and non-starchy) and limited fats.
  Interventions: Other: Standard low fat diet

INTERVENTIONS:
Other: Carbohydrate restricted group — Prescribed low carbohydrate diet with set recipes
  Arms: Carbohydrate restricted group
Other: Standard low fat diet — Diet with less than 20% total calorie intake from dietary fats
  Arms: Standard/Low fat diet group

SUMMARY:
Two-arm, parallel design with children between the ages of 10 - 18 with obesity and metabolic syndrome randomized (15 per group) to reduced-carbohydrate diet or a reduced-fat diet for 8 weeks.

DETAILED DESCRIPTION:
Two-arm, parallel design with participants randomized (15 per group) to reduced-carbohydrate diet or a reduced-fat diet for 8 weeks. Anthropometric evaluations, lab work for lipid levels, insulin and C peptide levels, resting energy expenditure evaluation, DXA scan and cardiovascular markers will occur at baseline during the initial clinic visit. Individual dietary counseling will be provided at baseline and as well as weekly diet-specific support will be provided with a phone call from the PI. Dietary intake will be assessed with weekly food records (weeks 1-8). The return visit on week 8 will include a visit identical to the initial visit except the resting energy expenditure will not be revaluated, and the participants will be asked to answer a questionnaire about the diet they were consuming.

ELIGIBILITY:
Inclusion Criteria: 3 out of 5 of the following criteria

* Metabolic syndrome with dyslipidemia
* (HDL <40mg/dL
* Triglyceride (TG) TG>150mg/dL)
* Glucose intolerance (fasting blood sugar >100mg/dL)
* Central adiposity (Waist circumference ≥90th percentile or adult cutoff if lower)
* Systolic BP ≥130 mm Hg or diastolic BP ≥85 mm Hg or treatment of previously diagnosed hypertension

Exclusion Criteria:

* Patient on medications known to induce dyslipidemia (systemic steroids, immunosuppressants)
* Pregnancy
* Untreated thyroid disease, heart disease, cancer, kidney disease
* Children on statin/fibrate treatments or other lipid-lowering medications
* Prior surgical procedure for weight control or current weight loss medication

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhuvana Sunil, MD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - Bhuvana Sunil, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carbohydrate Restricted Group | Standard/Low Fat Diet Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 12 (1) | 12 (1.3) | 12 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dyslipidemia Measures
Description: Baseline concentration of serum High-density Lipoprotein level in mg/dL
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
mg/dL | 30 (2) | 32 (2)

2. Primary Outcome: Dyslipidemia Measures
Description: Change in concentration of serum High density Lipoprotein in mg/dL
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL increase
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
mg/dL increase | 2 (0.5) | 2.3 (0.6)

3. Primary Outcome: Dyslipidemia Measures
Description: Baseline concentration of serum Triglyceride level in mg/dL
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
mg/dL | 160 (5.6) | 163 (2.6)

4. Primary Outcome: Dyslipidemia Measures
Description: Change in concentration of serum Triglyceride level in mg/dL
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
mg/dL | -8.7 (2.3) | -8.5 (2.1)

5. Primary Outcome: Dyslipidemia Measures
Description: Baseline concentration of serum lipoprotein particle number
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
nmol/L | 822 (125.6) | 821.6 (120.8)

6. Primary Outcome: Dyslipidemia Measures
Description: Change in concentration of serum lipoprotein particle number in percentage
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
percentage change | -0.052 (0.018) | -0.036 (0.016)

7. Primary Outcome: Dyslipidemia Measures
Description: Baseline concentration of serum lipoprotein particle concentration
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
mg/dL | 76.2 (8.36) | 77.1 (9.42)

8. Primary Outcome: Dyslipidemia Measures
Description: Change in concentration of serum lipoprotein particle concentration in percentage
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
percentage change | -0.062 (0.01) | -0.0617 (0.003)

9. Primary Outcome: Dyslipidemia Measures
Description: Baseline total serum high density lipoprotein particle number
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
micromol/L | 30.5 (1.8) | 30.62 (1.7)

10. Primary Outcome: Dyslipidemia Measures
Description: percentage Change in concentration of serum high density lipoprotein particle
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
percentage change | 02.76 (0.023) | 02.80 (0.051)

11. Primary Outcome: Dyslipidemia Measures
Description: Baseline concentration of serum small low-density lipoprotein particle concentration
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
nmol/L | 413.6 (18.3) | 418.2 (19.6)

12. Primary Outcome: Dyslipidemia Measures
Description: Percentage change in concentration of serum small low density lipoprotein particle
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
percentage change | -8.6 (0.58) | -8.15 (0.73)

13. Primary Outcome: Dyslipidemia Measures
Description: Baseline serum low-density lipoprotein size
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
nm | 21.62 (1.87) | 21.72 (2.1)

14. Primary Outcome: Dyslipidemia Measures
Description: Percentage change in concentration of serum small low-density lipoprotein size
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
percentage change | 1.65 (0.3) | 1.68 (0.24)

15. Primary Outcome: Insulin Resistance Indices
Description: Percentage change in Serum measure of Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
  HOMA_IR is a scale where a higher number means worse outcome
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
percentage change | -6.87 (0.38) | -7.65 (1.25)

16. Secondary Outcome: Insulin Resistance Indices
Description: Baseline Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
  HOMA_IR is a scale where a higher number means worse outcome
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: index score
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
index score | 2.15 (0.12) | 2.21 (0.16)

17. Secondary Outcome: Body Composition
Description: Dual-energy X-ray absorptiometry (DXA) - measure of body fat
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: % of total body weight
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
% of total body weight | 43.2 (5.8) | 45.6 (4.9)

18. Secondary Outcome: Body Composition
Description: Percent Change in Dual-energy X-ray absorptiometry (DXA) body fat
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
percentage change | -8.7 (2.1) | -8.84 (2.7)

19. Secondary Outcome: Surrogate Markers of Vascular Endothelial Function
Description: Baseline Pulse wave velocity
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
m/s | 11 (1) | 11.2 (1.6)

20. Secondary Outcome: Surrogate Markers of Vascular Endothelial Function
Description: Percentage Change in Pulse wave velocity
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
percentage change | -2 (1.5) | -2 (1.74)

21. Secondary Outcome: Surrogate Markers of Vascular Endothelial Function as Measured by Augmentation Index
Description: The Augmentation Index a measure of peripheral arterial stiffness
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
Percent | 81.8 (7.98) | 88.7 (8.76)

22. Secondary Outcome: Surrogate Markers of Vascular Endothelial Function as Measured by Augmentation Index
Description: The Augmentation Index a measure of peripheral arterial stiffness
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
Number analyzed (Participants) | 15 | 15
percentage change | -27 (1) | -28.6 (1.5)

ADVERSE EVENTS:
Time Frame: Each participant was assessed for adverse events during the duration of their participation for 8 weeks and additionally, for 8 weeks after their completion in the study for a total duration of 16 weeks from the time of enrollment in the study
Arm/Group | Standard/Low Fat Diet Group | Carbohydrate Restricted Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT03937960/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT03937960/SAP_001.pdf
  • Informed Consent Form (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT03937960/ICF_002.pdf